CLINICAL TRIAL: NCT01917253
Title: Standard Length Catheters vs Long Catheters in Peripheral Vein Cannulation. A Randomized Controlled Clinical Trial to Test the Complications.
Brief Title: Standard Length Catheters vs Long Catheters in Peripheral Vein Cannulation.
Acronym: Long&short
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASL TO2 Torino (Other)
Responsible Party: Principal Investigator, Tiziana De Prospo, Nurse, ASL TO2 Torino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 351/007A/2013
Record Dates: First submitted 2013-08-05; First posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Complications
Keywords: infiltration, phlebitis, occlusion, thrombosis
MeSH Terms: conditions — Phlebitis; Bites and Stings; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard length catheter (Experimental): Standard Device for peripheral vein cannulation
  Interventions: Device: Standard Device for peripheral vein cannulation
- Long catheter (Experimental): Standard Device for peripheral vein cannulation
  Interventions: Device: Long Catheters for peripheral vein cannulation

INTERVENTIONS:
Device: Standard Device for peripheral vein cannulation
  Arms: standard length catheter
Device: Long Catheters for peripheral vein cannulation
  Arms: Long catheter

SUMMARY:
The Long and Short is a prospective, randomized, controlled, open label trial to test the complications of different device for peripheral vein cannulation, standard length (about 5 cm in length) and long catheter (about 12 cm in length), inserted with Seldinger technique.

DETAILED DESCRIPTION:
The trial will compare the main complications: infiltration rate, phlebitis rate, occlusion and/or dislocation rate, thrombosis rate, number of percutaneous sticks, successful cannulation.

Will be made for a cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* infusional therapy more than 72 hours

Exclusion Criteria:

* need for central venous catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-09; Primary Completion 2013-10 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
complications rate | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Piero Riva, MD, Principal Investigator — ASLTO2- MECAU- Maria Vittoria Hospital
Locations (1):
- MECAU-Maria Vittoria Hospital, Torino, Torino, Italy